CLINICAL TRIAL: NCT01116271
Title: A Dose Finding and Phase II Study of Selumetinib (AZD6244) (Hyd-Sulfate) in Combination With Irinotecan, in 2nd Line Patients With K-ras or B-raf Mutation Positive Advanced or Metastatic Colorectal Cancer
Brief Title: Study of Selumetinib (AZD6244)(ARRY-142886) in Combination With Irinotecan in Previously Treated Patients With Colorec
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9010C00009; AGICC 09CRC02
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal; second line therapy; K-ras or B-raf mutations; response rate; Progression Free Survival
MeSH Terms: conditions — Colorectal Neoplasms | interventions — AZD 6244; Irinotecan

ARMS (1):
- 1 (Experimental): Selumetinib (AZD6244) in combination with irinotecan
  Interventions: Drug: AZD6244; Drug: Irinotecan

INTERVENTIONS:
Drug: AZD6244 — 50 or 75mg, capsules, PO, BID, 28 days
  Other Names: Selumetinib
Drug: Irinotecan — 180mg/m2, IV, Day 1& 15 of each cycle
  Other Names: Camptosar; Campto

SUMMARY:
The purpose of this study is to determine whether treatment with Selumetinib (AZD6244) (Hyd-Sulfate) in combination with Irinotecan as a second treatment in patients with K-ras or B-raf mutation will prevent tumor progression and prolong progression free survival.

DETAILED DESCRIPTION:
A Dose Finding and Phase II Study of Selumetinib (AZD6244) (Hyd-Sulfate) in Combination with Irinotecan, in 2nd Line Patients with K-ras or B-raf Mutation Positive Advanced or Metastatic Colorectal Cancer

ELIGIBILITY:
Inclusion Criteria:

- Histological or cytological confirmation of advanced or metastatic colorectal cancer with available tissue and tumor sample confirmed as K-ras or B-raf mutation positive. Current failure of 1st line anti-cancer therapy with an oxaliplatin and bevacizumab based regimen or patients relapsing within 12 months of completing adjuvant FOLFOX .

Exclusion Criteria:

- Treatment within 14 days prior to first study treatment with conventional therapy or treatment within 28 days prior to first study treatment with an investigational drug Prior treatment with a MEK or B-raf inhibitor or any irinotecan-containing regimen Prior treatment with a MEK or B-raf inhibitor or any irinotecan-containing regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Dose Finding will be calculated based upon toxicity screening and dose modification guidelines within protocol. | AEs will be assessed at each cycle visit, discontinuation treatment visit, and 30 days post last day of study treatment
Objective Response Rate will be assessed by the RECIST guideline documented in the European Journal of Cancer, 2009. | Tumor evaluation via RECIST guidelines will be done on screening visit, day 22 of every other cycle, and treatment discontinuation visit

SECONDARY OUTCOMES:
Safety of combination of Selumetinib (AZD6244) with irinotecan by SAE and AE documentation | AEs will be assesed at the screening visit, each cycle visit, treatment discontinuation date, and 30 days post last day of study treatment
PK of Selumetinib (AZD6244), N-desmethyl Selumetinib(AZD6244) and selumetinib (AZD6244) amide in combination with irinotecan | PK sample draws will take place on Day 1 and 15 of first cycle
Progression Free Survival (PFS) for patients with K-ras or B-raf mutations treated with combination of irinotecan and Selumetinib (AZD6244) | PFS will be determined via the RECIST guidelines on tumor measurement done on day 22 of every other cycle and on the treatment discontinuation visit

CONTACTS AND LOCATIONS:
Overall Officials: Howard Hochster, MD, Principal Investigator — Yale University; Lawrence Leichman, MD, Principal Investigator — Desert Regional Comprehensive Cancer Center
Locations (12):
- United States (12):
  - Research Site, Los Angeles, California
  - Research Site, Palm Springs, California
  - Research Site, Aurora, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Miami Beach, Florida
  - Research Site, New York, New York
  - Reserach Site, Chapel Hill, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Washington, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Seattle, Washington